CLINICAL TRIAL: NCT06030531
Title: Spasticity and Functional Recovery in Humans With Acute to Subacute Spinal Cord Injury.
Brief Title: Spasticity and Functional Recovery After SCI
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: Shirley Ryan AbilityLab (Other)
Responsible Party: Principal Investigator, Monica Perez, Principal Investigator, Shirley Ryan AbilityLab
Other Study IDs: STU00210582
Record Dates: First submitted 2022-04-07; First posted 2023-09-11 (Actual); Last update posted 2023-09-11 (Actual); Status verified 2023-09

CONDITIONS: Acute Spinal Cord Injury; Spinal Cord Injuries
Keywords: Spasticity; Recovery; Bio-markers
MeSH Terms: conditions — Spinal Cord Injuries; Muscle Spasticity

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — De-identified plasma and DNA extracts will be stored in key-lock secured -80 oC freezers in the Biologics Lab at SRALab until used for experimental purposes. Subjects will have the choice to allow researchers approved by this IRB to retain any leftover plasma or DNA extract taken during the study. These samples will be stored indefinitely and may be used only for IRB-approved research by IRB-approved researchers and personnel.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Inpatients: Prospective participants who meet the study inclusion criteria will be identified by bi-weekly chart review of all new admissions to the acute inpatient spinal cord injury unit at the Shirley Ryan AbilityLab (SRAlab).
  Eligible patients will be invited to participate by the clinical staff during their first week of admission.
  Interventions: Other: Measures of spasticity, connectivity and analysis of single nucleotide polymorphisms and biomarkers of inflammation; Other: Analysis of biomarkers
- Control group: We will enroll non-injured healthy individuals to compare the level of biomarkers
  Interventions: Other: Analysis of biomarkers

INTERVENTIONS:
Other: Measures of spasticity, connectivity and analysis of single nucleotide polymorphisms and biomarkers of inflammation — We will test for presence of biological markers in blood that may correlate with levels of spasticity or neurological recovery and functional improvement, including the presence or absence of neuroplastic genetic polymorphisms (e.g. BDNF Val66Met polymorphism), as well as circulating levels of neuroplastic(e.g. BDNF) or inflammatory factors (e.g. interleukins, TNF) that may affect neuronal growth and functional restoration.
  Groups: Inpatients
Other: Analysis of biomarkers — We will test for the presence of biological markers in the blood to compare the distribution of polymorphisms and biomarkers with the spinal cord injury patient population.

SUMMARY:
Spasticity is one of the most common symptoms manifested in humans with spinal cord injury (SCI). However, the neural mechanisms underlying the development of spasticity over time after an acute SCI are not yet understood. Using electrophysiological and imaging techniques along with traditional measurements of neurological recovery in the acute rehabilitation setting including physical exam and functional assessments; the investigators aim to examine the relationship between development of spasticity, residual descending motor pathways and functional and neurological recovery in humans with SCI from acute to subacute phase

DETAILED DESCRIPTION:
The purpose of this study is to measure changes to motor-evoked potentials (MEPs) and to evaluate if the development of spasticity is related to residual descending motor pathways and to a better neurological recovery and functional improvement in individuals with SCI from the acute to the subacute phase. The investigators will also test for the presence of biological markers in the blood that may correlate with levels of spasticity or neurological recovery and functional improvement, including the presence or absence of neuroplastic genetic polymorphisms (e.g. BDNF Val66Met polymorphism), as well as circulating levels of neuroplastic (e.g. BDNF) or inflammatory factors (e.g. interleukins, TNF) that may affect neuronal growth and functional restoration.

ELIGIBILITY:
Individuals with SCI:

Inclusion criteria:

* Male and females 18 years of age or greater
* Basic proficiency in English language communication
* Are admitted to the Shirley Ryan AbilityLab as a spinal cord injury patient
* International Standards for Neurological Classification of Spinal Cord Injury (ISNCSCI) level above L2
* American Spinal Cord Injury Association Impairment Scale (AIS) grades A, B, C, or D
* Patients with SCI within the first week of inpatient admission to the Shirley Ryan AbilityLab after sustaining a SC

Exclusion criteria:

* Under 18 years of age
* Severe cognitive impairment that precludes the ability to participate in a comprehensive physical exam or give verbal consent
* ISNCSCI level below L2
* People who have sustained SCI >30 days
* Uncontrolled medical problems including pulmonary, cardiovascular or orthopedic disease
* Any debilitating disease prior to the SCI that caused exercise intolerance
* Premorbid, ongoing major depression or psychosis, altered cognitive status
* History of head injury or stroke
* Vascular, traumatic, tumoral, infectious, or metabolic lesion of the brain, even without history of seizure, and without anticonvulsant medication
* History of seizures or epilepsy
* Ongoing cord compression or a syrinx in the spinal cord or people who suffer from a spinal cord disease such as spinal stenosis, spina bifida, MS, or herniated disk 13. Metal plate in skull
* Individuals with scalp shrapnel, cochlear implants, or aneurysm clips
* Skull fractures, skull deficits or concussion within the last 6 months
* Presence of orthoses and presence of spinal precautions or healing incisions that make the area inaccessible to the testing procedures. This criterion will be applied as needed for the specific study procedures that may need to access the areas under restriction.
* Formal diagnosis of Post-Traumatic Stress Disorder (PTSD)

Individuals in the control group:

Inclusion criteria:

1. Male and females 18 years of age or greater
2. Basic proficiency in English language communication

Exclusion criteria:

1. Under 18 years of age
2. Uncontrolled medical problems including pulmonary, cardiovascular, or orthopedic disease
3. History of neurological impairment or conditions affecting the Central Nervous System
4. Premorbid, ongoing major depression or psychosis, altered cognitive status
5. Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Prospective participants who meet the study inclusion criteria will be identified by bi-weekly chart review ofall new admissions to the acute inpatient spinal cord injury unit at the Shirley Ryan AbilityLab (SRAlab).Eligible patients will be invited to participate by the clinical staff during their first week of admission.
  Prospective participants that meet the inclusion criteria for the Control group will be recruited using various sources including the Shirley Ryan AbilityLab non-patient research database, participants who have taken part in our earlier studies, word of mouth, people who work at or visit our center and are interested in research participation.
Sampling Method: Non-Probability Sample
Enrollment: 240 (Estimated)
Dates: Start 2020-07-01 (Actual); Primary Completion 2023-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Modified Ashworth scale (MAS) | From the time of admission to the hospital and enrolled in the study till the time of discharge (up to 12 weeks)
  This clinical scale will be used by measuring resistance encountered during manual passive muscle stretching using a six-point ordinal scale (0=no increase in tone, 1/+1=slight increase in tone with a catch and release or minimal resistance at the end or less than half of the range of movement, respectively, 2=more marked increased tone through most of the range of movement but affected parts easily moved, 3=considerable increase in tone and passive movement difficultly, and 4=affected parts rigid)
Motor evoked potential (MEP) | From the time of admission to the hospital and enrolled in the study till the time of discharge (up to 12 weeks)
  Transcranial magnetic stimulation will be delivered and the coil will be positioned over the vertex and moved around this point to determine the optimal position for eliciting a motor evoked potentials (MEPs) in legs muscles.
First swing test (FST) | From the time of admission to the hospital and enrolled in the study till the time of the discharge (up to 12 weeks)
  We will use the pendulum test to measure muscle tone at the knee by using gravity to provoke muscle stretch reflexes during passive swinging of the lower limb.

SECONDARY OUTCOMES:
International Standards for Neurological Classification of Spinal Cord Injury (ISNCSCI) | From the time of admission to the hospital and enrolled in the study till the time of discharge (up to 12 weeks)
  At the time of the admission, after obtaining consent, and at the time of discharge, the chart will be reviewed to obtain the ISNCSCI score
Circulating biomarkers of inflammation and neuroplasticity | From the time of admission to the hospital and enrolled in the study till the time of discharge (up to 12 weeks)
  In this study, we will focus on tracking expression of key inflammatory cytokines that have been shown to play a pivotal role in activating the major nuclear factor kappa-B (NF-κB) inflammatory pathway. Specifically, we will characterize serum levels of pro-inflammatory cytokines interleukin-1 beta (IL-1β), interleukin-6 (IL-6), tumor necrosis factor (TNF-α) and anti-inflammatory marker interleukin-10 (IL-10). We will also measure levels of circulating neuroplasticity marker Brain-derived neurotrophic factor (BDNF)

CONTACTS AND LOCATIONS:
Overall Officials: Monica A Perez, PT, PhD, Principal Investigator — Shirley Ryan AbilityLab
Locations (1):
- Shirley Ryan AbilityLab, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: Undecided